CLINICAL TRIAL: NCT05672160
Title: CT Evaluated Sarcopenia Independently Predicts the Overal Survival After Transcatheter Aortic Valve Implantation
Brief Title: Overal Survival After TAVI According to Sarcopenia
Acronym: TAVI_Sarx
Status: Completed | Type: Observational
Sponsor: Nemocnice AGEL Trinec-Podlesi a.s. (Other)
Responsible Party: Principal Investigator, Matej Pekar, MD, PhD, Mr. Matej Pekar, MD, PhD, Nemocnice AGEL Trinec-Podlesi a.s.
Other Study IDs: TAVI_Sarx
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Sarcopenia; Aortic Valve Stenosis
Keywords: sarcopenia; survival; TAVI
MeSH Terms: conditions — Sarcopenia; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT evaluated sarcopenia — At L3 level of CT scan we will measure the area and density of muscles and fat tissue. We devided the patients to sarcopenia and non-sarcopenia groups according to these values.

SUMMARY:
The goal of this observational study is to compare the overal survival after transcatheter aortic valve implantation (TAVI) according to sarcopenia status evaluated from preprocedural CT scans.

The main question it aims to answer is:

• Is CT evaluated sarcopenia an independent predictor of overal survival after TAVI?

DETAILED DESCRIPTION:
The patients suffering from aortic valve stenosis, that are not eligible for cardiosurgery were indicated to miniinvasive transcatheter aortic valve implantation (TAVI). The follow up of 930 patients were done in time interval from 1 to 11 years. In every patient the preprocedural CT scans were done. From these CT scans the L3 cross sections will be used for sarcopenia evaluation. Then we will statisticaly evaluate the overal survival after TAVI procedure in the relation with sarcopenia status. We will answer the main question: Is CT evaluated sarcopenia an independent predictor of overal survival after TAVI?

ELIGIBILITY:
Inclusion Criteria:

* patients udergone TAVI procedure

Exclusion Criteria:

* patients with incomplete TAVI procedure, patients without clinical follow up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients indicated for TAVI procedure because of the critical aortic valve stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 930 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Overal survival | 11 years
  Time from the TAVI procedure to death

CONTACTS AND LOCATIONS:
Locations (1):
- AGELTrinecPodlesi, Třinec, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: Undecided